CLINICAL TRIAL: NCT03059394
Title: Validation of Manual Muscle Testing and the Myositis Activity Profile Assessments in Patients With Inflammatory Myositis
Brief Title: Validation of Rehab Assessments in Myositis Patients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0022
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Myositis
Keywords: reliability; validity; measurement error
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Non intervention study — Test - Retest of measurements
  Other Names: Test retest study

SUMMARY:
The aim of the study is to evaluate the psychometric properties (content and construct validity, reliability, measurements error, as well as possible floor and ceiling effects) of both the assessments MMT8 and the myositis activity profile in patients with IM.

DETAILED DESCRIPTION:
This study evaluates the validity and reliability of two health related instruments that assess disease relevant functions and disabilities in patients with IM: the manual muscle testing 8 (MMT8) and the myositis activity profile (MAP). This study is needed to determine the psychometric properties of these two assessments. Provided that both the MMT8 and the MAP show good psychometric properties, these assessments could be used in the rehabilitation process and intervention programs of patients with IM to determine progress in muscle strength and activity in daily life.

Methodology: Reliability (Test re-test study and validity (cross sectional study) of a short form of MMT 8 and a questionnaire to assess difficulties in activities of daily life (MAP) in myositis patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of polymyositis or dermatomyositis or inflammatory myositis associated disorders (e.g. Scleroderma, Systematic lupus erythematosus, Sjögren's syndrome)
* Age over 18
* Sufficiently understanding of German language
* able to understand and follow verbal and written instructions
* signed informed consent to participate in the study

Exclusion Criteria:

* Diagnosis of inclusion body myositis
* Pulmonary hypertension
* Osteoporosis
* Severe cardiovascular and/or pulmonary disease
* Pain syndrome
* Paresis

Inclusion Criteria aged and gender matched healthy controls (Systematic lupus erythematosus, Sjögren's syndrome)

* Age over 18
* Sufficiently understanding of German language
* able to understand and follow verbal and written instructions
* signed informed consent to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Patients with diagnosed inflammatory myopathy
  2. Age and gender matched controls
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Manual Muscle Testing 8 (MMT8) | 15 minutes
  The strength of 8 Muscle groups is tested in a defined position and rewarded with a score varying from 0 (No visible movement) to 10 (holds test position against strong pressure) and summed for a potential score from 0-80.

SECONDARY OUTCOMES:
Quantitative Muscle Testing | 15 Minutes
  Hand Held Dynamometer in Newton
Functional Index 2 | 30 minutes
  Evaluates muscle endurance of the upper & lower extremity and neck flexors movements: amount of repetitions.
Functional Test Battery (FTB): Test 1 Self-Performed Physical Performance Test. | Total FTB: 1 1/4 hours
  Time in seconds to get up and sit down 5 times from a chair.
Functional Test Battery (FTB): Balance Test | Total FTB: 1 1/4 hours
  Time in seconds (max 10 sec.) 1) balance feet together, 2) semi-tandem, 3) full-tandem stand.
Functional Test Battery ( FTB): Walk test ( 4 m) | Total FTB: 1 1/4 hours
  Time in sec.
Functional Test Battery ( FTB): 1 leg stand | Total FTB: 1 1/4 hours
  Time in sec.
Functional Test Battery ( FTB): Grip ability Test | Total FTB: 1 1/4 hours
  Time in sec. (max 60 sec.)
Functional Test Battery ( FTB): Jamar grip test | Total FTB: 1 1/4 hours
  Strength in Kg.
Functional Test Battery ( FTB): Pile Test | Total FTB: 1 1/4 hours
  Work = Joule & Performance = Watt
Functional Test Battery ( FTB): 6 Minute walk-test | Total FTB: 1 1/4 hours
  Meters during 6 minutes
Modified Myositis Activity Profile | 30 Minutes
  34 item Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Baschung Pfister Pierrette, MPH, Study Chair — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The dataset analyzed in the current study is available from the corresponding author(s) on reasonable request.